CLINICAL TRIAL: NCT01209754
Title: HIV Prevention Agent Pregnancy Exposure Registry: EMBRACE Study
Brief Title: EMBRACE (Evaluation of Maternal and Baby Outcome Registry After Chemoprophylactic Exposure)
Acronym: EMBRACE
Status: Completed | Type: Observational
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: MTN-016; 3UM1AI068633 (NIH); 10737 (Other Grant/Funding Number: DAIDS Protocol ID)
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Chemoprophylactic Exposure; Mother; Infant; malformations; HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pregnant Women: Pregnant women exposed to an HIV prevention study agent during pregnancy
- Infant: Infants resulting from pregnancies where there exists maternal HIV prevention agent exposure

SUMMARY:
The Prevention Agent Pregnancy Exposure Registry, also known as EMBRACE (Evaluation of Maternal and Baby Outcome Registry After Chemoprophylactic Exposure) is a prospective observational cohort investigation of exposures to study agents under investigation for HIV prevention. The study population will consist of female participants who are identified as becoming pregnant during their participation in a microbicide or PrEP trial, or who have had planned exposures in pregnancy safety studies as well as their babies resulting from these pregnancies. This study will only enroll babies who have not yet reached their 1 year birth date.

DETAILED DESCRIPTION:
The Prevention Agent Pregnancy Exposure Registry, also known as EMBRACE (Evaluation of Maternal and Baby Outcome Registry After Chemoprophylactic Exposure) is a prospective observational cohort study of maternal exposures to investigational HIV prevention agents. Approximately 550 pregnant participants and 400 live infants will be offered enrollment. The study population will consist of current or recent female participants identified as becoming pregnant during microbicide or PrEP trials, or who have had planned exposures in pregnancy safety studies. This study will also include infants resulting from those pregnancies. This protocol will monitor for adverse pregnancy and delivery outcomes, monitor the prevalence of major malformations, evaluate growth parameters of infants during the first year of life, and evaluate the prevalence and persistence of HIV drug resistance mutations in a cohort of infants who were either exposed to active study agents or not exposed to active study agents while in utero.

ELIGIBILITY:
Inclusion Criteria: Mother cohort

1. Able and willing to provide written informed consent to take part in the study
2. During participation in a parent protocol, has/had a known confirmed pregnancy, meeting at least one of the following sets of criteria in A or B:

   A. Two consecutive monthly study visits, at least 14 days apart, with positive pregnancy tests, in the absence of signs/symptoms of miscarriage or participant report of pregnancy termination.

   B. One or more of the following assessments:
   * Auscultation of fetal heart tones
   * Positive pregnancy test confirmed by clinic staff in the presence of clinically confirmed enlarged uterus
   * Positive pregnancy test confirmed by clinic staff in the presence of missed menses (no menses occurring at least 60 days from the first day of the last menses) by participant report (For amenorrheic or irregularly cycling women, two consecutive positive hCG tests (criterion A) or any of the other clinical signs of pregnancy included under the criteria B listing will be used to confirm MTN-016 eligibility).
   * Clinical assessment of fetal movement
   * Demonstration of pregnancy by ultrasound
3. Able and willing to provide adequate locator information, as defined in site SOPs

Note: Participants do not have to be currently enrolled or engaged in follow-up in a parent protocol to participate in EMBRACE.

Inclusion Criteria: Infant cohort

1. Has written informed consent provided by parent(s)/guardian to take part in the study in a manner consistent with local standards, site Institutional Review Board (IRB) guidance and the US Code of Federal Regulations (CFR)
2. Born to EMBRACE participant mother from pregnancy concurrent with participation in parent study

Exclusion Criteria: Mother cohort

1. Has any condition that in the opinion of the investigator or designee, would complicate interpretation of study outcome data, make participation in the study unsafe, or otherwise interfere with achieving the study objectives
2. Pregnancy outcome occurred greater than one year ago

Exclusion Criteria: Infant cohort

1. Has any condition that, in the opinion of the investigator or designee, would complicate interpretation of study outcome data, make participation in the study unsafe, or otherwise interfere with achieving the study objectives
2. Has reached 1 year birth date

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of female participants who become or became pregnant during HIV prevention agent trials, or who have or had planned exposures in pregnancy safety studies, and the infants resulting from those pregnancies. Mother participants must still be pregnant, or have had a pregnancy outcome diagnosis less than one year before screening/enrollment, and infant participants must be less than one year old. The study may include HIV-uninfected and -infected participants. Mothers may participate in EMBRACE without participation of their infants; however, infants whose mothers have not enrolled in EMBRACE will not participate.
Sampling Method: Non-Probability Sample
Enrollment: 873 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy and delivery outcomes comparison | Duration of Study
  To compare adverse pregnancy and delivery outcomes between participant mothers assigned to an active agent with those of mothers assigned to placebo/control. Pregnancy and delivery outcomes of interest are:
  * delivery prior to 37 completed weeks of gestation
  * stillbirth or intrauterine fetal demise (≥ 20 weeks)
  * spontaneous abortion (< 20 weeks)
  * ectopic pregnancy
  * intrapartum hemorrhage
  * postpartum hemorrhage
  * non-reassuring fetal status
  * chorioamnionitis
  * hypertensive disorders of pregnancy
  * gestational diabetes
  * intrauterine growth restriction
Major malformations comparison | Duration of Study
  To compare the prevalence of major malformations identified in the first year of life between infants of mothers assigned to an active agent with those of infants of mothers assigned to placebo/control. Major malformations are defined as structural abnormalities with surgical, medical, or cosmetic importance.

SECONDARY OUTCOMES:
Infant growth parameters comparison | Duration of Study
  To compare growth parameters in the first year of life between infants of mothers assigned to an active agent with those of mothers assigned to placebo/control. Growth parameters of interest are weight, length, and head circumference at birth, one month, six months and 12 months.
HIV drug resistance mutations comparison | Duration of Study
  2. To evaluate the prevalence and persistence of HIV drug resistance mutations in plasma among HIV-infected infants.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beigi, MD, Study Chair — Microbicide Trials Network
Locations (17):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- South Africa (11):
  - Wits Reproductive Health Institute (WRHI), Johannesburg, Gauteng
  - CAPRISA-The Aurum Institute, Johannesburg, Guateng
  - CAPRISA eThekwini, Durban, KwaZulu-Natal
  - Perinatal HIV Research Unit (PHRU), Johannesburg, Soweto
  - South African MRC HIV CTU Med Research Council; Botha's Hill Clinical Research Site, Durban
  - South African MRC HIV CTU Med Research Council; Isipingo, Durban
  - South African MRC HIV CTU Med Research Council; Overport, Durban
  - South African MRC HIV CTU Med Research Council; R.K. Khan Hospital, Durban
  - South African MRC HIV CTU Med Research Council; Tongaat, Durban
  - South African MRC HIV CTU Med Research Council; Umkomaas, Durban
  - South African MRC HIV CTU Med Research Council; Verulam, Durban
- Makerere University-Johns Hopkins University Collaboration, Kampala, Uganda
- Zimbabwe (3):
  - UZ-UCSF HIV Prevention Trials Unit, Chitungwiza, Seke South
  - UZ-UCSF HIV Prevention Trials Unit, Harare, Spilhaus
  - UZ-UCSF HIV Prevention Trials Unit, Chitungwiza, Zengeza

REFERENCES:
- [Result] Makanani B, Balkus JE, Jiao Y, Noguchi LM, Palanee-Phillips T, Mbilizi Y, Moodley J, Kintu K, Reddy K, Kabwigu S, Jeenariain N, Harkoo I, Mgodi N, Piper J, Rees H, Scheckter R, Beigi R, Baeten JM. Pregnancy and Infant Outcomes Among Women Using the Dapivirine Vaginal Ring in Early Pregnancy. J Acquir Immune Defic Syndr. 2018 Dec 15;79(5):566-572. doi: 10.1097/QAI.0000000000001861. PMID 30383589
- [Result] Mhlanga FG, Noguchi L, Balkus JE, Kabwigu S, Scheckter R, Piper J, Watts H, O'Rourke C, Torjesen K, Brown ER, Hillier SL, Beigi R. Implementation of a prospective pregnancy registry for antiretroviral based HIV prevention trials. HIV Clin Trials. 2018 Feb;19(1):8-14. doi: 10.1080/15284336.2017.1411419. Epub 2017 Dec 21. PMID 29268654